CLINICAL TRIAL: NCT02016508
Title: Intravitreal Injection of Human Bone Marrow Derived Mesenchymal Stem Cell in Patients With Dry Age-related Macular Degeneration(AMD)
Brief Title: Safety Study of Use of Autologous Bone Marrow Derived Stem Cell in Treatment of Age Related Macular Degeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Collaborators: Hassan , Hosny , M.D. M.Sc (Unknown); Samour , Hany M.D. M.Sc (Unknown); Ismail , Mahmoud M.D. M.Sc (Unknown); Higazy , Hasan M.D. M.Sc (Unknown); Abou el kheir, Wael, M.D. M.Sc. (Unknown); Gabr, Hala , M.D. M.Sc. (Unknown); Bakry, Sayed , phD. M.Sc. (Unknown)
Responsible Party: Principal Investigator, abdelhakim mohamed safwat, assistant lecturer ophthalmology department al-azhar university, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT 4619792013; 4619792013 (Other Grant/Funding Number: Al-Azhar university)
Record Dates: First submitted 2013-05-18; First posted 2013-12-20 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Age Related Macular Degeneration
Keywords: Adult bone marrow stem cells; AMD
MeSH Terms: conditions — Macular Degeneration

ARMS (1):
- autologous bone marrow stem cells (Experimental): use of autologous bone marrow derived stem cells as intravitreal injection in AMD patients
  Interventions: Drug: autologous bone marrow derived stem cells

INTERVENTIONS:
Drug: autologous bone marrow derived stem cells — intravitreal injection of autologous bone marrow stem cells in 0.1 ml volume

SUMMARY:
The purpose of this Phase I/II study is to investigate the safety and preliminary efficacy of unilateral intravitreally transplantation of adult bone marrow stem cells in subjects with geographic atrophy secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
This study is an open-label investigation of the safety and preliminary efficacy of unilateral intravitreal injection of autologous bone marrow stem cells in subjects with Geographic Atrophy secondary to Age-Related Macular Degeneration (AMD). Subjects will be enrolled based on specific inclusion/exclusion criteria and evaluated at regular post transplant intervals.

Human central nervous system -stem cells will be transplanted by a vitreoretinal surgeon. The transplantation will be conducted in the eye with the inferior best-corrected visual acuity (BCVA) (i.e., the Study Eye). Only the Study Eye will undergo transplantation. The adult bone marrow stem cells will be administered into the vitreous cavity through a standard surgical approach.

Moxifloxacin 300 mg(once per day ) will be administered orally to all subjects for a period of five days ( 2 days pre and post operatively) .

Subjects will be monitored frequently for a total of one year after adult bone marrow stem cells cell injection .

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration with geographic atrophy (GA)
* Only patients with a specific degree and extent of GA will be eligible
* Subjects with best-corrected visual acuity (BCVA) of less than or equal to 20/400 in the Study Eye
* No prior or current choroidal neovascularization in either eye
* Able to provide written informed consent prior to any study related procedures
* Agree to comply in good faith with all conditions of the study and to attend all required study visits

Exclusion Criteria:

* Prior vitreal or retinal surgery in the previous 6 months
* Glaucoma
* Atrophic macular disease of any other cause
* Diabetic retinopathy or diabetic macular edema in either eye
* Previous organ, tissue or bone marrow transplantation
* Autoimmune disease
* Allergy to moxifloxacin
* Current or prior malignancy (or is on chemotherapy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
number of subjects with adverse events | 6 months
  Descriptive analysis of frequency and types of adverse events experienced by each subject during the study period

SECONDARY OUTCOMES:
Assessment of visual function changes from the base line | 6 months
  assessment will include Change in the mean of BCVA, Optical Coherence Tomography imaging, fluorescein angiography, slitlamp examination with fundus photography, Electroretinographic evidence (mfERG) showing enhanced activity in the location

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university medical school (Benin-cairo) ophthalmology department, Cairo, Nasr City, Egypt